CLINICAL TRIAL: NCT06187285
Title: Efficay and Safety of Empagliflozin Versus Sitagliptin for the In-patient Management of Hyperglycemia: Randomised Control
Brief Title: Efficay and Safety of Empagliflozin Versus Sitagliptin for the In-patient Management of Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medanta, The Medicity, India (Other)
Collaborators: Diabetes & Endocrinology Foundation (Unknown)
Responsible Party: Principal Investigator, Dr Mohammad Shafi Kuchay, Senior Consultant, Medanta, The Medicity, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMDNB01
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin 25 mg (Experimental)
  Interventions: Drug: Empagliflozin 25 MG
- Sitagliptin 100 mg (Active Comparator)
  Interventions: Drug: Sitagliptin 100mg

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Patient will get Empagliflozin 25
  Arms: Empagliflozin 25 mg
Drug: Sitagliptin 100mg — Patient will get Sitagliptin 100 mg
  Arms: Sitagliptin 100 mg

SUMMARY:
Clinical guidelines from professional organizations have recommended the use of multidose insulin regimens as the preferred therapy for glycaemic control in patients admitted to hospital in a non-intensive-careunit setting. The use of a basal-bolus regimen with a once daily basal insulin and rapid-acting insulin analogs before meals has been shown to improve glycaemic control and to reduce the rate of hospital complications in general medical and surgical patients with type 2 diabetes.The basal-bolus regimen however is labour intensive, requiring several insulin injections, and is associated with a high risk of hypoglycaemia. Hypoglycaemia has been reported in 12% to 32% of patients in general medicine and surgery with type 2 diabetes treated with basal-bolus insulin regimens.Because of these limitations, alternative treatment regimens are needed that could improve glycaemic control and clinical outcomes, while facilitating care and minimising the risk of hypoglycaemia in patients with diabetes.

DETAILED DESCRIPTION:
The management of hyperglycemia in noncritically ill, hospitalized patients with diabetes mellitus is mainly based on insulin therapy . This usually consists of one dose of long-acting basal insulin and three doses of rapid-acting premeal bolus insulins (basal-bolus insulin). Basal-bolus insulin therapy is, however, labor intensive, requiring multiple insulin injections per day and multiple daily blood glucose checks. The use of oral antidiabetic medications has generally not been recommended for patients admitted to the hospital. This is because of the lack of safety and efficacy . data, and concerns about hypoglycemia. Oral medication usually has a slow onset of action that might preclude daily dose adjustments and have considerable interactions with concomitantly administered drugs. Oral antidiabetic medications are also withheld during hospitalization because of several safety concerns related to altered pharmacokinetics in cases of end-stage organ disease, such as renal or liver failure. Dipeptidyl peptidase-4 inhibitors (sitagliptin and linagliptin) have been studied for the treatment of hospitalized patients in the noncritical care setting. Complementary to insulin therapy, these drugs improved glycemia and were found to be safe. Sodium-glucose cotransporter type 2 (SGLT2) inhibitors are another class of oral glucose-lowering medication that is increasingly being used in patients with T2D, due to multiple pleiotropic efects . These drugs reduce cardiovascular mortality, especially by reducing the risk of heart failure, and also improve renal outcomes . Recently, two randomized controlled trials demonstrated improvement in several cardiac outcomes when SGLT2 inhibitors (empaglifozin and dapaglifozin) were initiated in patients admitted for acute heart failure, with or without diabetes .This trial aimed to examine the efficacy and safety of Empagliflozin in Hopitalised patients in comparison to Sitagliptin.

Hyperglycaemia is a common and serious health-care problem in hospitals, reported in approximately 30% of patients in general medicine and surgery with and without a history of previous diabetes mellitus..Extensive evidence from observational and randomised clinical studies in patients admitted to hospital indicates that hyperglycaemia, in patients both with and without diabetes, is a predictor of poor outcome.In such patients, hyperglycaemia is associated with prolonged hospital stay, increased incidence of infections, hospital complications, and death. Improvement in glycaemic control with insulin therapy has been shown to reduce the risk of infection and complications in patients in hospital critical-care units and in patients admitted to general surgical and medical services. Although insulin therapy is the standard of care in hospitals, it is a source of medication errors and increased risk of hypoglycemia. An analysis of medication errors between 2006 and 2008 revealed that insulin was the drug with the greatest number of medication errors in hospitals. Hypoglycemia in the hospital has been associated with adverse cardiovascular outcomes such as prolonged QT intervals, ischemic electrocardiogram changes/angina, arrhythmias, sudden death, and increased inflammation..In addition, insulin-induced hypoglycemia is associated with increases in C-reactive protein and proinflammatory cytokines (TNF-α, interleukin-1β, IL-6, and interleukin-8), markers of lipid peroxidation, ROS, and leukocytosis.. The use of oral antidiabetic agents is not recommended in hospitals because few data are available regarding their safety and efficacy in the inpatient setting. Major limitations to the use of oral agents in the hospital include their side effect profiles and slow onset of action, which does not allow for rapid attainment of glycemic control or dose adjustments to meet the changing needs of acutely ill patients. Sodium glucose co-transporter 2 (SGLT-2) inhibitors are a new class of oral antidiabetic medications that increase urinary glucose excretion by reducing renal glucose reabsorption in the proximal convoluted tubules. Canaglifozin and dapaglifozin are the two available drugs approved by the U.S. Food and Drug Administration for management of type 2 diabetes. Both agents are effective in reducing A1C by ~ 0.6-0.8%, with a low risk of hypoglycemia. A recently published, randomized pilot study assessed the safety and efficacy of SGLT2 inhibitor Dapagliflozin for the inpatient management of type 2 diabetes(37). In this study done in hospitalized patients with T2D admitted for cardiac surgery, treatment with dapaglifozin 10 mg once a day plus basal-bolus insulin or basal-bolus insulin regimen alone in the early postoperative period resulted in similar glycemic control. There was a rapid improvement in glycemic control in both groups, without signifcant diferences in mean daily blood glucose, number and percentage of blood glucose values within the target of 70-180 mg/dL, total daily insulin doses and number of daily insulin injections. As the use of dapaglifozin complementary to basal-bolus insulin did not reduce insulin dose or the number of insulin injections per day, therefore dapaglifozin lacks glycemic efficacy in hospitalized cardiac surgery patients. A recently published, randomized pilot study assessed the safety and efficacy of the DPP-4 inhibitor sitagliptin for the inpatient management of type 2 diabetes(31).In this trial, patients treated with diet, oral antidiabetic agents, or a low daily insulin dose (≤ 0.4 units/kg/day) were randomized to sitagliptin alone or in combination with low-dose insulin glargine or to a basal-bolus insulin regimen plus supplemental doses of insulin lispro. Glycemic control improved similarly in all treatment groups. The trial met the non-inferiority threshold for the primary endpoint of differences between the sitagliptin-basal and basal-bolus groups for mean daily blood glucose concentrations. Of patients with type 2 diabetes admitted to general medicine and surgery services in hospital, treatment with a daily dose of sitagliptin and basal insulin or with a basal bolus regimen resulted in similar glycaemic control and frequency of complications.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18-years and above with type 2 diabetes and a random blood glucose concentration of 140-400 mg/dL who were being treated with diet or oral antidiabetic drugs or had a total daily insulin dose of 0•6 units per kg or less, admitted to general medicine or surgery

Exclusion Criteria:

Patients with a blood glucose concentration greater than 400mg/dL or with current or previous history of diabetic ketoacidosis,

Type 1 diabetes,

Hyperglycaemia without a known history of diabetes

Patients expected to be without oral intake for more than 48 h

Patients admitted to or expected to require admission to an intensive care unit

Clinically relevant hepatic disease or impaired renal function [eGFR] <30 mL/min per 1•73 m²)

Pregnancy, and any mental health condition rendering the patient unable to give informed consent

Current or recurrent uti(more than 2 times in last 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Mean blood glucose concentration | The first 7 days of therapy in hospital
  Blood glucose will be measured pre-breakfast, pre-lunch, pre-dinner and bed time. Mean daily blood glucose concentration will be calculated to determine differences in inpatient glycemic control in patients with type 2 diabetes treated with empagliflozin 25 mg (Empa Group) or sitagliptin 100 mg (Sita Group). Both groups will receive basal insulin and/or supplemental bolus insulin

SECONDARY OUTCOMES:
Number of basic glucose readings between 70 mg/dl and 180 mg/dl before meals and bed time in hospitalized patients | The first 7 days of therapy in hospital
Number of hypoglycemic episodes (BG < 70 mg/dl and 54 mg/dl) in hospitalized patients. | The first 7 days of therapy in hospital
Number of severe hypoglycemia (< 54 mg/dl) episodes in hospitalized patients | The first 7 days of therapy in hospital
Number of episodes of severe hyperglycemia (BG > 240 mg/dl) in hospitalized patients. | The first 7 days of therapy in hospital
Daily dose of basal insulin, daily dose of prandial insulin, and total daily dose in hospitalized patients. | The first 7 days of therapy in hospital
Hospital complications | The first 7 days of therapy in hospital
ketonemia | The first 7 days of therapy in hospital
Diabetic acidosis | The first 7 days of therapy in hospital
Glycated hemoglobin | The first 7 days of therapy in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Division Of Endocrinology & Diabetes, Medanta The Medicity, Gurgaon, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Umpierrez GE, Isaacs SD, Bazargan N, You X, Thaler LM, Kitabchi AE. Hyperglycemia: an independent marker of in-hospital mortality in patients with undiagnosed diabetes. J Clin Endocrinol Metab. 2002 Mar;87(3):978-82. doi: 10.1210/jcem.87.3.8341. PMID 11889147
- [Background] Moghissi ES, Korytkowski MT, DiNardo M, Einhorn D, Hellman R, Hirsch IB, Inzucchi SE, Ismail-Beigi F, Kirkman MS, Umpierrez GE; American Association of Clinical Endocrinologists; American Diabetes Association. American Association of Clinical Endocrinologists and American Diabetes Association consensus statement on inpatient glycemic control. Diabetes Care. 2009 Jun;32(6):1119-31. doi: 10.2337/dc09-9029. Epub 2009 May 8. No abstract available. PMID 19429873
- [Background] Umpierrez GE, Hellman R, Korytkowski MT, Kosiborod M, Maynard GA, Montori VM, Seley JJ, Van den Berghe G; Endocrine Society. Management of hyperglycemia in hospitalized patients in non-critical care setting: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2012 Jan;97(1):16-38. doi: 10.1210/jc.2011-2098. PMID 22223765
- [Background] Pomposelli JJ, Baxter JK 3rd, Babineau TJ, Pomfret EA, Driscoll DF, Forse RA, Bistrian BR. Early postoperative glucose control predicts nosocomial infection rate in diabetic patients. JPEN J Parenter Enteral Nutr. 1998 Mar-Apr;22(2):77-81. doi: 10.1177/014860719802200277. PMID 9527963
- [Background] Capes SE, Hunt D, Malmberg K, Pathak P, Gerstein HC. Stress hyperglycemia and prognosis of stroke in nondiabetic and diabetic patients: a systematic overview. Stroke. 2001 Oct;32(10):2426-32. doi: 10.1161/hs1001.096194. PMID 11588337
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168
- [Background] Williams LS, Rotich J, Qi R, Fineberg N, Espay A, Bruno A, Fineberg SE, Tierney WR. Effects of admission hyperglycemia on mortality and costs in acute ischemic stroke. Neurology. 2002 Jul 9;59(1):67-71. doi: 10.1212/wnl.59.1.67. PMID 12105309
- [Background] Kuchay MS, Khatana P, Mishra M, Surendran P, Kaur P, Wasir JS, Gill HK, Singh A, Jain R, Kohli C, Bakshi G, Radhika V, Saheer S, Singh MK, Mishra SK. Dapagliflozin for inpatient hyperglycemia in cardiac surgery patients with type 2 diabetes: randomised controlled trial (Dapa-Hospital trial). Acta Diabetol. 2023 Nov;60(11):1481-1490. doi: 10.1007/s00592-023-02138-4. Epub 2023 Jun 29. PMID 37380728
- [Background] Kuchay MS, Mishra SK, Mehta Y. Empagliflozin induced euglycemic diabetic ketoacidosis in a patient undergoing coronary artery bypass graft despite discontinuation of the drug 48 hours prior to the surgery. Diabetes Metab Syndr. 2021 May-Jun;15(3):909-911. doi: 10.1016/j.dsx.2021.04.016. Epub 2021 Apr 22. No abstract available. PMID 33915345
- [Background] Pasquel FJ, Gianchandani R, Rubin DJ, Dungan KM, Anzola I, Gomez PC, Peng L, Hodish I, Bodnar T, Wesorick D, Balakrishnan V, Osei K, Umpierrez GE. Efficacy of sitagliptin for the hospital management of general medicine and surgery patients with type 2 diabetes (Sita-Hospital): a multicentre, prospective, open-label, non-inferiority randomised trial. Lancet Diabetes Endocrinol. 2017 Feb;5(2):125-133. doi: 10.1016/S2213-8587(16)30402-8. Epub 2016 Dec 8. PMID 27964837